CLINICAL TRIAL: NCT06994546
Title: Intra Articular Hyaluronic Acid (ArtiBest ® ) for Knee Osteoarthritis: A Post-market, Open Label, Long Term Study
Brief Title: ArtiBest for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBI-AB-202408
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthristis
Keywords: hyaluronic acid; intra articular injection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AB (Experimental)
  Interventions: Device: ArtiBest ® Intra articular Injection

INTERVENTIONS:
Device: ArtiBest ® Intra articular Injection — single intra articular injection of 3 ml (one syringe) per knee joint. Each syringe contains 20 mg/mL sodium hyaluronate.

SUMMARY:
The goal of this clinical trial is to evaluate the real-world effectiveness and safety of ArtiBest in the treatment of knee osteoarthritis. The main questions it aims to answer are:

1. The change from baseline The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score at 26 weeks post injection.
2. The change from baseline VAS resting pain score at 12 and 26 weeks post injection.
3. The change from baseline The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score at 12 weeks post injection.
4. The change from baseline Patient's Global Assessment PGA) using VAS scoring at 12 and 26 weeks post injection.
5. The OMERACT OARSI responder rate at 12 and 26 weeks post injection.
6. The VAS satisfaction score at 12 and 26 weeks post injection
7. The incidence of Adverse events reported during the study period.

Participants will undergo a single injection of ArtiBest at treatment visit, and three follow up visits at week 4 , 12 , and 26.

DETAILED DESCRIPTION:
This single center, single arm, open label, interventional study aims to assess the effectiveness and the safety profiles of ArtiBest ® Intra articular Injection(MAXIGEN BIOTECH INC., Taiwan). It plans to enroll approximately 60 eligible patients to receive a 3 ml single pre-filled syringe per knee joint at the treatment visit. Each syringe contains 20 mg/mL sodium hyaluronate. Follow-up visits will be at 4 weeks(a telephone contact by the investigator), 12 weeks and 26 weeks after the injections. All endpoints are planning to evaluate the change between baseline(pre-treatment) and 12 and 26 weeks post-injection. The OMERACT-OARSI responder rate will also be calculated. And the exploratory endpoints will evaluate the change in the range of motion (ROM) at 12 and 26 weeks post-injection. Additionally, the Kellgren-Lawrence grade (KL grade) at baseline and 26 weeks, as well as the target joint space at baseline and 26weeks, will also be analyzed. In general, the change from the baseline of continuous data will be performed by paired t-test or Wilcoxon signed-rank test. The statistical analysis for primary endpoint will be one-sided under a significance level of 0.025. Unless otherwise specified, other statistical analysis will be two-sided under a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age from 35 to 85 years.
* Subject with x ray imaging evidence of knee OA as Kellgren Lawrence grade = 2 or 3 within 1 month at screening.
* Subject diagnosed with mild to moderate knee OA, particularly in patients who failed to respond adequately to conservative nonpharmacologic therapies or analgesics.
* Subject with a 100 mm VAS resting pain score ≥ 30 mm in the studied knee at both the screening and treatment visit (screening visit and treatment visit can be on the same day)
* Able and willing to comply with all study visits and procedures.
* Willin g and capable of providing written informed consent.

Exclusion Criteria:

* Subjects with known hypersensitivity to hyaluronate.
* Subjects with infections or skin diseases in the area of the injection site.
* Pregnancy or breast feeding woman.
* Joining other interventional trial s within 3 months prior to injecting this study product
* Subject receive an intra articular (IA) injection of Hyaluronic Acid (HA) and/or steroid in target knee within 6 months prior to the trial
* Subjects with rheumatoid arthritis
* Any surgery to the target knee within the 12 months prior to the trial, or surgery to the contralateral knee or other weight bearing joint if it will interfere with knee assessments

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The change of The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score | Week 0 and 26 weeks post injection
  The change from baseline The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score at 26 weeks post injection.

SECONDARY OUTCOMES:
The change of VAS resting pain score | Week 0, 12 and 26 weeks post injection
  The change from baseline VAS resting pain score at 12 and 26 weeks post injection.
The change of The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score | Week 0, 12 weeks post injection
  The change from baseline The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score at 12 weeks post injection.
The change of Patient's Global Assessment (PGA) | Week 0, 12 and 26 weeks post injection
  The change from baseline Patient's Global Assessment (PGA) using VAS scoring at 12 and 26 weeks post injection.
The OMERACT OARSI responder rate | 12 and 26 weeks post injection
  The OMERACT OARSI responder rate at 12 and 26 weeks post injection.
The VAS satisfaction score | 12 and 26 weeks post injection
  The VAS satisfaction score at 12 and 26 week s post injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan